CLINICAL TRIAL: NCT02307383
Title: Pilot Study of the Effectiveness of Probiotics and Lactitol for the Intestinal Decolonization of People Carriers of Klebsiella Pneumoniae Producers of Carbapenemase OXA-48-type: DesProbiOXA Study
Brief Title: Pilot Study of the Effectiveness of Probiotics and Lactitol for the Decolonization of OXA-48 (Carbapenemase) Producing Klebsiella Pneumoniae Among Rectal Carriers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Desprobioxa
Record Dates: First submitted 2014-11-20; First posted 2014-12-04 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Bacterial Colonization
Keywords: SDD (Selective Digestive Decolonization); OXA 48; carbapenemase; probiotics
MeSH Terms: interventions — lactitol; Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactitol and Lactobacillus (Experimental): Lactitol monohydrated 10g (Emportal®), 1 sachet dissolved in water, three times a day for 21 days.
  Lactobacillus acidophilus, 1 x 109 UFC and Lactobacillus Biphidus 1 x 109 UFC, (Infloran Berna), 2 tablets by mouth, three times a day for 21 days.
  Interventions: Drug: Lactitol; Drug: Lactobacillus

INTERVENTIONS:
Drug: Lactitol
  Other Names: Emportal
Drug: Lactobacillus
  Other Names: Infloran Berna

SUMMARY:
The combination of Lactitol and Probiotics (Lactobacillus acidophilus and Lactobacillus Biphidus) administered orally is an effective strategy of intestinal decolonization of Enterobacter produced OXA-48-type carbapenemase.

The purpose of this study is to determine the effectiveness of Lactitol and Probiotics for the intestinal decolonization of people who carried Klebsiella pneumoniae produced OXA-48-type Carbapenemase.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Have signed the informed consent to participate.
* Have evidence of intestinal colonization by KP-OXA-48 during the period of screening.
* Start of intestinal colonization by KP-OXA-48, > 6 months of starting treatment.
* Absence of exclusion criteria

Exclusion Criteria:

* Be hospitalized for an acute process at the time of inclusion.
* Take antibiotics (oral , intramuscular or intravenous ) at the time of inclusion.
* Having diarrhea in the two weeks prior to the inclusion.
* Baseline electrolyte abnormalities requiring supplementation : Hypokalemia (K <3 mEq / L), hypomagnesemia (Mg <1.8 mEq / L ), hypocalcemia (Ca < 8mg/dL )
* Suffering from digestive diseases : Crohn's disease, ulcerative colitis , celiac disease, irritable bowel syndrome , intestinal resection, colostomies.
* Neutropenia ( neutrophil count < 1.00 x 10 3 / uL ) or other situations of severe immunosuppression , including continued use of systemic steroids (at least 1mg/kg/day of prednisone or equivalent for more than 1 month) and other forms of pharmacological immunosuppression deemed by the investigator.
* Diabetes mellitus poorly controlled ( HgA1c > 8 mmol / mol ).
* Taking antisecretory inhibitors, proton pump or anti -H2.
* Advanced chronic renal failure (GFR < 30 ml / min)
* Being a carrier of endovascular prosthetic devices, including long-term central catheters.
* Having significant valvulopathy on the opinion of the investigator.
* Surgical intervention of gastrointestinal tract in the last three months.
* Treatment with systemic corticosteroids or immunosuppressive.
* Allergy or intolerance to lactose or lactitol or Infloran .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the combination of lactitol and probiotics, administered orally to achieve intestinal decolonization of KP-OXA-48 in people. | Six weeks

SECONDARY OUTCOMES:
Evaluate the effectiveness of lactitol and probiotics administered orally for intestinal decolonization of KPOXA -48 in people. | Three weeks and six weeks
  In people at the time of the end of treatment (End of treatment Response) and 3 weeks after end of treatment (Short-term response).
Evaluate the safety and tolerability of the combination of lactitol and probiotics (Lactobacillus acidophilus and Bifidobacterium bifidum ) measured by the increase of diarrhea, flatulence, abdominal pain, loss of appetite and weight loss | Three weeks
Analyze the effect of the combination of lactitol and probiotics (Lactobacillus acidophilus and Bifidobacterium bifidum ) administered orally on intestinal microbiota of carriers of KP- OXA -48 | Three weeks
Evaluate the time from the start of treatment with lactitol and probiotics (Lactobacillus acidophilus and Bifidobacterium bifidum ) to intestinal decolonization in those patients who achieved sustained response. | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Arnalich, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- [Derived] Ramos-Ramos JC, Lazaro-Perona F, Arribas JR, Garcia-Rodriguez J, Mingorance J, Ruiz-Carrascoso G, Borobia AM, Pano-Pardo JR, Herruzo R, Arnalich F. Proof-of-concept trial of the combination of lactitol with Bifidobacterium bifidum and Lactobacillus acidophilus for the eradication of intestinal OXA-48-producing Enterobacteriaceae. Gut Pathog. 2020 Apr 7;12:15. doi: 10.1186/s13099-020-00354-9. eCollection 2020. PMID 32280375
- See also: Related Info — http://www.idipaz.es/